CLINICAL TRIAL: NCT04028596
Title: StudY of Effect of Nimodipine and Acetaminophen on Postictal Symptoms After ECT
Brief Title: Measuring Blood Flow in the Brain After Epileptic Activity
Acronym: SYNAPSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: University of Twente (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NL68690.091.18
Record Dates: First submitted 2019-07-08; First posted 2019-07-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Epilepsy; Depression; Postictal Delirium; Electroconvulsive Therapy
Keywords: Epilepsy; Depression; Electroconvulsive Therapy; Postictal; Clinical Trial; Postictal hypoperfusion/hypoxia
MeSH Terms: conditions — Epilepsy; Depression; Hypoxia | interventions — Acetaminophen; Nimodipine

STUDY DESIGN:
Intervention Model Description: This study makes use of a 3 x 3 crossover design, in which patients receive a randomized sequence of interventions in pairs of 3 (acetaminophen, nimodipine, no intervention), with a maximum of 12 interventions/measurements.
Who Masked: Investigator
Masking Description: The PROBE design will be used in this study, in which the principal investigator will be blinded to the administration of drugs until the end of the study. The other principal investigator will know about administration, but will not be involved in testing patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acetaminophen (Active Comparator): Trade name: Paracetamol Pharmaceutical form: Tablet (oral use) Once 1000 mg 2h before the ECT-session. Total maximum of five times over the course of weeks
  Interventions: Drug: Paracetamol
- Nimodipine (Active Comparator): Trade name: Nimotop Pharmaceutical form: Film-coated tablet (oral use) Once 60mg 2h before the ECT-session. Total maximum of five times over the course of weeks.
  Interventions: Drug: Nimotop
- Control (No Intervention): Glass of water (50cc) only. Once 2h before the ECT-session. Total maximum of five times over the course of weeks.

INTERVENTIONS:
Drug: Paracetamol — once, 1000mg, 2 h before ECT session
  Other Names: RVG 107336
  Arms: Acetaminophen
Drug: Nimotop — once, 60mg, 2 h before ECT session
  Other Names: RVG 12060
  Arms: Nimodipine

SUMMARY:
In this clinical trial, postictal phenomena (i.e., headache, delirium) will be investigated after administration of acetaminophen and nimodipine in depressed patients receiving electroconvulsive therapy (ECT). Postictal phenomena are thought to result from decreased cerebral blood flow and decreased oxygen concentration in the brain. It is expected that acetaminophen and nimodipine will reduce these postictal phenomena, compared to no treatment, because they target these mechanisms.

DETAILED DESCRIPTION:
Postictal phenomena, such as sensory, motor or memory deficits, headache, delirium, and psychosis, are common manifestations after electroconvulsive therapy (ECT) induced seizures. Also, postictal phenomena add to the burden of seizures in patients with epilepsy. The pathophysiology of these phenomena is poorly understood and effective treatments are not available (Fisher RS, 2000; Krauss & Theodore, 2010). Recently, seizure-induced postictal vasoconstriction with cerebral hypoperfusion was observed in experimentally induced seizures in rats. Treatment with acetaminophen or calcium antagonists decreased hypoperfusion and postictal phenomena (Farrell, 2016, 2017).

The objective of this research is to study the effect of acetaminophen and nimodipine to reduce postictal phenomena after ECT induced seizures.

A prospective, three conditions crossover trial will be conducted, with randomized condition allocation, open-label treatment, and blinded end-point evaluation (PROBE design; Hansson, Hedner, & Dahlof, 1992).

Thirty-three adult (age >17 years) patients referred to treatment with ECT for a depressive episode will be included to achieve a statistical power of .80. This will be feasible in one year.

A single dose of nimodipine (60 mg) or acetaminophen (1000 mg) or no additional treatment will be given prior to a maximum of 12 ECT-sessions per patient. Patients will be randomly assigned to predefined treatment sequences. EEG and MRI measures will serve as main outcome measures, as well as psychometric tests.

Data will be stored on two separate hard disks, one including patient sensitive information for identification, the other with anonymized data only (for the sponsor).

Patients will be recruited by doctors at Rijnstate Hospital Arnhem. A mixed model with repeated measurements analysis will be conducted for the primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Adulthood (age > 17 years);
* Current clinical diagnosis of depressive episode (unipolar, bipolar, schizoaffective);
* Willingness and ability to give written informed consent and willingness and ability to understand, to participate and to comply with the study requirements.

Exclusion Criteria:

* Known adverse or allergic reactions to acetaminophen or nimodipine;
* Chronic use of acetaminophen, calcium-antagonists or NSAID's that cannot be interrupted for less than two days before the ECT-session;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Time to EEG normalization | Change from ictal to baseline EEG activity, up to 12 times per patient (across 6 weeks)
  quantitative metric of EEG background evolution over time, in seconds (will be assessed at baseline, during electroconvulsive therapy, and immediately afterwards for approximately 1 hour)

SECONDARY OUTCOMES:
Postictal reorientation time (by Sobin, 1995) | immediately after each ECT session, up to 12 times per patient (across 6 weeks)
  Five questions regarding reorientation will be asked in an interval of 5 minutes after electroconvulsive shock therapy has ended. If the patient can answer 4 out of the 5 questions correctly, this is determined as the final score (in minutes). The scale ranges from 5 to 100 minutes. These scores indicate the time frame a patient needs until he/she is fully conscious and reoriented. Higher values indicate that a patient needs more time to regain reorientation.
Structural MRI | baseline, in the first hour after 3 electroconvulsive therapy sessions, after approx. 3 months, after approx. 6 months, lasts approx. 5 min.
  Isovoxel T1-weighted data (to make volumetric changes); is part of the MRI sequence (takes in total approximately 25 minutes)
Arterial Spin Labeling MRI | baseline, in the first hour after 3 electroconvulsive therapy sessions, after approx. 3 months, after approx. 6 months, lasts approx. 7 min.
  measures cerebral perfusion levels
Resting state functional MRI | baseline, in the first hour after 3 electroconvulsive therapy sessions, after approx. 3 months, after approx. 6 months, lasts approx. 5 min.
  used for brain mapping, measures functional organization (and connectivity) of certain brain areas
Diffusion Tensor Imaging | baseline, in the first hour after 3 electroconvulsive therapy sessions, after approx. 3 months, after approx. 6 months, lasts approx. 5 min.
  measures diffusion in the brain to estimate the axonal organization of the brain

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen A van Waarde, MD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The EEG, MRI, and psychometric data will be shared with the University of Twente and the Amsterdam UMC. All patient data will be anonymized so that it cannot be connected to the patients. Demographic data will also be included in these files and anonymized.
Supporting Information: CSR, Analytic Code
Time Frame: Data will be archived for 15 years (according to the standard practice of Rijnstate Hospital). Data will become available as of the last date of testing (approx. December 2020).
Access Criteria: Data will be shared with experienced data analysts at the Amsterdam UMC (MRI analyses).

REFERENCES:
- [Background] Farrell JS, Gaxiola-Valdez I, Wolff MD, David LS, Dika HI, Geeraert BL, Rachel Wang X, Singh S, Spanswick SC, Dunn JF, Antle MC, Federico P, Teskey GC. Postictal behavioural impairments are due to a severe prolonged hypoperfusion/hypoxia event that is COX-2 dependent. Elife. 2016 Nov 22;5:e19352. doi: 10.7554/eLife.19352. PMID 27874832
- [Background] Farrell JS, Colangeli R, Wolff MD, Wall AK, Phillips TJ, George A, Federico P, Teskey GC. Postictal hypoperfusion/hypoxia provides the foundation for a unified theory of seizure-induced brain abnormalities and behavioral dysfunction. Epilepsia. 2017 Sep;58(9):1493-1501. doi: 10.1111/epi.13827. Epub 2017 Jun 20. PMID 28632329
- [Background] Fisher RS, Schachter SC. The postictal state: a neglected entity in the management of epilepsy. Epilepsy Behav. 2000 Feb;1(1):52-9. doi: 10.1006/ebeh.2000.0023. PMID 12609127
- [Background] Hansson L, Hedner T, Dahlof B. Prospective randomized open blinded end-point (PROBE) study. A novel design for intervention trials. Prospective Randomized Open Blinded End-Point. Blood Press. 1992 Aug;1(2):113-9. doi: 10.3109/08037059209077502. PMID 1366259
- [Background] Krauss G, Theodore WH. Treatment strategies in the postictal state. Epilepsy Behav. 2010 Oct;19(2):188-90. doi: 10.1016/j.yebeh.2010.06.030. Epub 2010 Aug 17. PMID 20719574
- [Background] Sobin C, Sackeim HA, Prudic J, Devanand DP, Moody BJ, McElhiney MC. Predictors of retrograde amnesia following ECT. Am J Psychiatry. 1995 Jul;152(7):995-1001. doi: 10.1176/ajp.152.7.995. PMID 7793470
- [Derived] Pottkamper JCM, Verdijk JPAJ, Stuiver S, Doesschate FT, van Putten MJAM, Hofmeijer J, van Waarde JA, van Wingen GA. Postictal resting-state connectivity changes after electroconvulsive therapy-induced seizures. Eur Arch Psychiatry Clin Neurosci. 2025 Jul 14. doi: 10.1007/s00406-025-02043-7. Online ahead of print. PMID 40659830
- [Derived] Verdijk JPAJ, Pottkamper JCM, Verwijk E, van Wingen GA, van Putten MJAM, Hofmeijer J, van Waarde JA. Study of effect of nimodipine and acetaminophen on postictal symptoms in depressed patients after electroconvulsive therapy (SYNAPSE). Trials. 2022 Apr 18;23(1):324. doi: 10.1186/s13063-022-06206-y. PMID 35436940